CLINICAL TRIAL: NCT04100759
Title: Pharmacokinetics and Pharmacodynamics of Sildenafil in Adult Smokers and Non-smokers
Brief Title: A Comparative Pharmacokinetic and Pharmacodynamic Study of Sildenafil in Adult Smokers and Non Smokers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Drug Research Centre, Cairo, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Raslan, QC Manager and Clinical pharmacy Msc student, Drug Research Centre, Cairo, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIL-RES-0119
Record Dates: First submitted 2019-09-12; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Erectile Dysfunction; Smoking; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Erectile Dysfunction; Smoking | interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-Smokers (Experimental): Subjects administer one tablet of sildenafil 50 mg
  Interventions: Drug: Sildenafil 50 mg Oral Tablet
- Cigarette Smokers (Experimental): Subjects administer one tablet of sildenafil 50mg
  Interventions: Drug: Sildenafil 50 mg Oral Tablet
- Cannabis Smokers (Experimental): Subjects administer one tablet of sildenafil 50mg
  Interventions: Drug: Sildenafil 50 mg Oral Tablet

INTERVENTIONS:
Drug: Sildenafil 50 mg Oral Tablet — Sildenafil 50 mg Oral Tablet
  Other Names: Viagra 50 mg film coated tablets

SUMMARY:
Smokers are at higher risk of developing Erectile dysfunction (ED) independent of age and comorbidities. Sildenafil is a cytochrome p3A4 (CYP3A4) substrate used for enhancing the erectile function in males. The study purpose is to determine the effect of smoking on male sexual function based on the international index of erectile function score (IIEF) and investigate the effect of smoking (Cigarettes or marijuana) on the pharmacokinetics and pharmacodynamics of sildenafil.

DETAILED DESCRIPTION:
The study is a randomized, single dose, one way, open label, parallel study in thirty-six (36) subjects randomized into three groups;group(1) included twelve(12) healthy non-smoker males, group(2) included twelve(12) healthy smokers (Cigarettes) and group(3) included twelve(12) healthy smokers (marijuana).

Each group received a single dose of Viagra 50 mg film coated tablet (Sildenafil 50 mg) Blood samples were collected at the following sampling intervals: pre-dose administration, 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8,10, 12 and 24 hours post dose.

Blood samples were centrifuged and plasma was separated and stored at -80 degree Celsius till time of analysis.

Plasma concentrations of sildenafil were determined by liquid chromatography tandem mass spectrometry (LC/MS/MS)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age 18-55 years.
* Ideal weight with ideal body mass index(BMI).
* Non-contributory history and normal physiological examination.
* Laboratory data within normal limits.
* Performance and compliance.
* The subjects should be without known history of alcohol or drug abuse problems
* Subjects who are cigarette smokers
* Subjects who are cannabis smokers
* Subjects who are non-smokers

Exclusion Criteria:

* A known hypersensitivity to the drug.
* Gastrointestinal diseases.
* Auto immune diseases.
* Renal diseases or dysfunction.
* Cardiovascular disease of any type.
* Pancreatic disease including diabetes.
* Hepatic disease.
* Hematological, osteopathic, or pulmonary disease.
* History of alcoholism or drug abuse.
* Serious Psychological illness.
* Positive HIV.
* Abnormal (out of range) laboratory values.
* Subject who have taken any medication less than two weeks of the trials starting date.
* Subject who have donated blood or who have been in multiple dosing studies requiring a large volume of blood (more than 500 ml) to be drawn within six weeks preceding the start of the trials.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — subjects are to provide their national IDs to confirm that subjects are male subjects
Enrollment: 36 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration in plasma (Cmax) | up to 3 hours post-dose
  Maximum drug concentration in plasma measured in nano-grams per milliliters (ng/ml)
Area under the plasma concentration-time curve from time zero to the last quantifiable concentration post-dose (AUC0→t) | up to 24 hours post-dose
  Area under the plasma concentration-time curve from time 0 to time(t) measured in nano-grams multiplied by hours and divided by milliliters (ng.h/ml)

SECONDARY OUTCOMES:
Time to Maximum drug concentration in plasma (tmax) | up to 3 hours post-dose
  Time corresponding to maximum drug concentration in plasma measured in Hours(h)
Elimination half life of drug in plasma ( t½) | Up to 24 hours post-dose
  Elimination half life of drug measured in Hours(hr)
Area under the plasma concentration-time curve from time 0 to infinity | Up to 24 hours post-dose
  Area under the plasma concentration-time curve from time 0 to infinity measured in nano-grams multiplied by hours and divided by milliliters (ng.h/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A Sabri, phD, Principal Investigator — Ainshams university; Mohammed M Hussein, Msc student, Principal Investigator — Ainshams university; Mohamed A Raslan, Study Director — Drug Research Centre, Cairo, Egypt
Locations (1):
- Drug Research Centre, Cairo, Sheraton Heliopolis, Egypt